CLINICAL TRIAL: NCT05674513
Title: Disparities in Emergency Contraceptive Metabolism Dictate Efficacy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Edelman, Professor, OB/GYN, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 24952; 1R01HD105866-01A1 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2023-01-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Contraceptive Usage
Keywords: Ulipristal acetate; Emergency contraception
MeSH Terms: conditions — Contraception Behavior | interventions — ulipristal acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active CYP3A5 Allele (Active Comparator): Ulipristal acetate 30mg orally x 1 dose with pharmacokinetic and pharmacodynamics testing in individuals with active CYP3A5 alleles
  Interventions: Drug: Ulipristal acetate
- Inactive CYP3A5 Allele (Active Comparator): Ulipristal acetate 30mg orally x 1 dose with pharmacokinetic and pharmacodynamics testing in individuals without active CYP3A5 alleles
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate — Evaluating the pharmacodynamic and pharmacokinetic outcomes after 1 dose of Ulipristal acetate 30mg in individuals with and without active CYP3A5 alleles

SUMMARY:
The purpose of this study is to learn more about why some people are at greater risk for oral emergency contraceptive failure while others are not. The investigators want to learn if genetic differences impact the risk of emergency contraception failure.

DETAILED DESCRIPTION:
Each of us can respond differently to a drug or medication based on our genetics. An emergency contraceptive, ulipristal acetate or UPA, normally works by stopping or delaying the ovary from releasing an egg (ovulation). Our bodies break down UPA in order to use it through a system call the cytochrome P450 pathway but this pathway can be faster or slower depending on our genetics. The investigators want to learn more about how our individual genetic differences in this pathway change how the ovary responds to UPA. The overall goal of this research is to improve the effectiveness of emergency contraception for all people.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women
* Aged 18-40
* regular menses (every 21-35 days) experiencing ovulatory cycles proven by a single progesterone level of 3 ng/mL or greater during the luteal phase of the screening cycle.

Exclusion Criteria:

* Pregnant, seeking pregnancy, or breastfeeding
* Known allergy to study medication
* Recent use of hormonal contraception
* Irregular periods (<21 days or >35 day cycles)
* Routine use of nonsteroidal anti-inflammatory drugs
* Metabolic disorders
* Smoking
* Any condition that would preclude the provision of informed consent
* Using drugs (within 2 weeks of study enrollment) known to interfere with the metabolism of UPA as well as drugs known to be CYP3A4 inducers, inhibitors, or CYP3A drug substrates

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Delay in follicular rupture | over 1 menstrual cycle (assessed up to approximately 30 days)
  Follicular rupture (yes/no) by ultrasound. Defined as the disappearance of or >50% reduction in size of the leading follicle
Concentration of UPA | 5 days after taking study drug
  mean concentration maximum (Cmax) for UPA

CONTACTS AND LOCATIONS:
Overall Officials: ALISON EDELMAN, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States